CLINICAL TRIAL: NCT04652063
Title: Using Osteopathic Manipulative Medicine on Preterm Infants in the Neonatal Intensive Care Unit to Reduce Neuromotor Developmental Delays
Brief Title: Osteopathic Manipulative Medicine to Reduce Developmental Delays
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Ronnie Guillet, Professor of Pediatrics (Neonatology), University of Rochester
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Study00005304
Record Dates: First submitted 2020-11-25; First posted 2020-12-03 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Extreme Prematurity; Neurodevelopmental Abnormality
Keywords: osteopathic manipulative medicine (OMM); test of infant motor performance (TIMP); neurodevelopmental outcomes

STUDY DESIGN:
Intervention Model Description: Randomization 1:1 to control and intervention group
Who Masked: Care Provider, Outcomes Assessor
Masking Description: The individual performing the developmental assessment will be unaware of study arm assignment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- OMM (Experimental): Neonates randomized to receive osteopathic manipulation
  Interventions: Other: Osteopathic Manipulative Medicine
- Control (No Intervention): Neonates randomized to receive standard care only

INTERVENTIONS:
Other: Osteopathic Manipulative Medicine — Osteopathic evaluation and treatment (gentle touch according to published protocols) will take about 15 - 20 minutes, and will be performed every 7 - 10 days during the infant's NICU stay once they reach at minimum of at least 28 weeks corrected gestational age and until they reach 36 weeks corrected gestational age.
  Arms: OMM

SUMMARY:
This randomized clinical trial seeks to determine if osteopathic manipulative medicine (OMM) increases the likelihood of improved neurodevelopmental outcomes as estimated by the Test of Infant Motor Performance (TIMP).

DETAILED DESCRIPTION:
Hypothesis: High risk preterm infants born <34 weeks of gestation who receive OMM, compared to the standard supportive care, will have improved neuromotor development scores on the TIMP.

Specific Aims and Objectives:

Primary aim: To determine the difference in TIMP scores between infants who receive OMM and those who receive only standard neonatal intensive care unit (NICU) care.

Secondary aims:

* To compare length of stay between infants who receive OMM and those who receive only standard NICU care.
* To compare growth parameters including weight, length, and head circumference, (both means and Z scores) prior to discharge between infants who receive OMM and those who receive only standard NICU care.
* To compare percentage of subjects requiring nasogastric, orogastric, or gastrostomy tube feeds at discharge between infants who receive OMM and those who receive only standard NICU care.

ELIGIBILITY:
Inclusion Criteria:

* 23 0/7- 33 6/7 weeks' gestational age (GA) at birth, ≥28 0/7 weeks' GA at time of consent
* stable enough to tolerate gentle manipulation

Exclusion Criteria:

* > 33 6/7 weeks' GA at birth
* known congenital and genetic abnormalities affecting neurodevelopment
* known conditions requiring surgical intervention
* severe intracranial hemorrhage or other severe neurologic complications
* parents unable to read and understand English

Ages: 1 Day to 14 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 150 (Actual)
Dates: Start 2021-01-05 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2023-07-30 (Actual)

PRIMARY OUTCOMES:
Test of Infant Motor Performance (TIMP) | At approximately 36 weeks' corrected gestational age
  Standardized, validated assessment of risk for developmental delay; expected range: 20 - 90 with higher scores indicating less risk for developmental delay

SECONDARY OUTCOMES:
Length of stay | At NICU discharge, assessed up to 1 year
  Number of days in Neonatal Intensive Care Unit (NICU)
Growth parameters - weight | at 36 weeks' corrected gestational age and discharge
  weight z-score
Growth parameters - length | at 36 weeks' corrected gestational age and discharge
  length z-score
Growth parameters - head circumference | at 36 weeks' corrected gestational age and discharge
  head circumference z-score
Need for nasogastric (NG), orogastric (OG), or gastrostomy tube feeds at discharge | at NICU discharge, assessed up to 1 year
  Number of neonates requiring NG, OG, or gastrostomy feeds at discharge from NICU

CONTACTS AND LOCATIONS:
Overall Officials: Ronnie Guillet, MD, PhD, Principal Investigator — University of Rochester
Locations (2):
- United States (2):
  - Golisano Children's Hospital, Rochester, New York
  - University of Rochester, Rochester, New York

IPD SHARING:
Plan to Share IPD: No
No plans to share HPI and data for individual participants at this time.

REFERENCES:
- [Background] Cerritelli F, Martelli M, Renzetti C, Pizzolorusso G, Cozzolino V, Barlafante G. Introducing an osteopathic approach into neonatology ward: the NE-O model. Chiropr Man Therap. 2014 May 9;22:18. doi: 10.1186/2045-709X-22-18. eCollection 2014. PMID 24904746
- [Background] Wang L, He JL, Zhang XH. The efficacy of massage on preterm infants: a meta-analysis. Am J Perinatol. 2013 Oct;30(9):731-8. doi: 10.1055/s-0032-1332801. Epub 2013 Jan 15. PMID 23322391
- [Background] Cerritelli F, Pizzolorusso G, Renzetti C, Cozzolino V, D'Orazio M, Lupacchini M, Marinelli B, Accorsi A, Lucci C, Lancellotti J, Ballabio S, Castelli C, Molteni D, Besana R, Tubaldi L, Perri FP, Fusilli P, D'Incecco C, Barlafante G. A multicenter, randomized, controlled trial of osteopathic manipulative treatment on preterms. PLoS One. 2015 May 14;10(5):e0127370. doi: 10.1371/journal.pone.0127370. eCollection 2015. PMID 25974071
- [Background] Campbell SK, Swanlund A, Smith E, Liao PJ, Zawacki L. Validity of the TIMPSI for estimating concurrent performance on the test of infant motor performance. Pediatr Phys Ther. 2008 Spring;20(1):3-10. doi: 10.1097/PEP.0b013e31815f66a6. PMID 18300928